CLINICAL TRIAL: NCT06659393
Title: Entresto Tablets and Granules for Pediatric Specified Drug-use Survey (Pediatric Chronic Heart Failure, CLCZ696F1401)
Brief Title: Entresto Tablets and Granules for Pediatric Specified Drug-use Survey (Pediatric Chronic Heart Failure)
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696F1401
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is multicenter, single-arm, non-interventional, centrally enrolled specified drug-use survey to investigate the safety of Entresto Tablets or Entresto Granules for Pediatric in pediatric patients with chronic heart failure in actual clinical settings for up to 52 weeks after administration.

DETAILED DESCRIPTION:
This specified drug-use survey is conducted to collect information on the safety specifications of Entresto in pediatric patients with chronic heart failure in Japan in actual clinical settings, and to investigate the occurrence of events related to the safety specifications, the risk factors associated with these events, and the status of Entresto administration including the accidental administration of capsule-shaped container (Granules for Pediatric). The subjects of this study are pediatric patients and a long-term observation of 1 year (52 weeks) has been set.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent by a legally acceptable representative must be obtained before the start of treatment with Entresto.
2. Patients who received Entresto for the first time under the indication of chronic heart failure
3. Pediatric patients aged 1 to < 18 years old at the start of treatment with Entresto

Exclusion criteria

1. Patients who have received drugs containing the same ingredient as Entresto (including investigational products and drugs for post-marketing clinical study)
2. Patients for whom Entresto is contraindicated according to the package insert

   * Patients with a history of hypersensitivity to any ingredients of Entresto
   * Patients currently under treatment with angiotensin-converting enzyme inhibitors or within 36 hours of discontinuation of treatment with angiotensin-converting enzyme inhibitors (alacepril, imidapril hydrochloride, enalapril maleate, captopril, quinapril hydrochloride, cilazapril hydrate, temocapril hydrochloride, delapril hydrochloride, trandolapril, benazepril hydrochloride, perindopril erbumine, lisinopril hydrate).
   * Patients with a history of angioedema (including angioedema due to angiotensin II receptor blockers or angiotensin-converting enzyme inhibitors, hereditary angioedema, acquired angioedema, and idiopathic angioedema etc.)
   * Patients with diabetes mellitus under treatment with aliskiren fumarate (excluding patients with markedly poorly controlled blood pressure despite other antihypertensive therapies)
   * Patients with severe hepatic impairment (Child-Pugh class C)
   * Pregnant women or women who may be pregnant

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Japanese pediatric patients with chronic heart failure using Entresto Tablets and Granules
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of events related to hypotension, hyperkalemia, renal impairment/renal failure, and dehydration | one year
  To confirm the occurrence status up to 52 weeks of events related to hypotension, hyperkalemia, renal impairment/renal failure, and dehydration as safety specifications of Entresto administration in pediatric patients with chronic heart failure in actual clinical settings.

SECONDARY OUTCOMES:
Occurrence of events related to hypotension, hyperkalemia, renal impairment/renal failure, and dehydration by the risk factors | one year
  To investigate the impact of risk factors on the occurrence of hypotension, hyperkalemia, renal impairment/renal failure, and dehydration as safety specifications.
Occurrence of the accidental administration of the capsule-shaped container (Granules for Pediatric) | one year
  To confirm the occurrence status of the accidental administration of the capsule-shaped container (Granules for Pediatric).
Occurrence of adverse events, SAEs, adverse drug reactions, and serious adverse drug reactions | one year
  To confirm the occurrence of adverse events, SAEs, adverse drug reactions, and serious adverse drug reactions.
Administration status of Entresto during the observation period | one year
  To confirm the administration status of Entresto used in actual clinical settings.

CONTACTS AND LOCATIONS:
Locations (25):
- Japan (25):
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Ōmura, Nagasaki
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Hidaka, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Kumamoto

IPD SHARING:
Plan to Share IPD: No